CLINICAL TRIAL: NCT01652534
Title: Efficacy of Amantadine for Gait Dysfunction and Gait Freezing in Patients With Parkinson's Disease
Brief Title: Efficacy Study of Amantadine to Treat Gait Dysfunction and Freezing in Parkinson's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to lack of recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Tanya Simuni, Professor of Neurology Director, Parkinson's Disease and Movement Disorders Center, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: M012010
Record Dates: First submitted 2011-08-15; First posted 2012-07-30 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Freezing of gait; gait dysfunction
MeSH Terms: conditions — Parkinson Disease | interventions — Amantadine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amantadine (Active Comparator): Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day
  Interventions: Drug: Amantadine
- placebo (Placebo Comparator): Sugar Pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine — Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day. Amantadine will then be administered orally twice daily in the morning with breakfast and at noon with lunch (AM and NN).
  Other Names: Symmetrel
  Arms: Amantadine
Drug: Placebo — Sugar Pill
  Other Names: Sugar Pill
  Arms: placebo

SUMMARY:
The purpose of this study is to explore the efficacy of the drug Amantadine for the treatment of freezing of gait in patients with Parkinson's Disease. The investigators hypothesize that amantadine is useful for management of freezing of gait in subjects with Parkinson's Disease.

DETAILED DESCRIPTION:
Subjects who meet the eligibility requirements for the study will be randomized to Amantadine versus a matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with idiopathic PD as determined by UK brain bank diagnostic criteria
2. H&Y stage 2.5-3
3. Presence of freezing of gait (FOG) as determined by UPDRS Part I score > 2
4. Ability to walk for 2 minutes in the ON and OFF state
5. Stable regimen of PD medications for 30 days prior to screening
6. Ability to comply with the study procedures
7. If female, be either post menopausal for at least 2 years, surgically sterilized or have undergone hysterectomy or, if of child bearing potential they must be willing to avoid pregnancy by using an adequate method of contraception as defined in Section 6.4.10 for four weeks prior to, during and four weeks after the last dose of trial medication. For the purposes of this trial, women of childbearing potential are defined as all female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive.
8. Willing and able to provide informed consent.

Exclusion Criteria:

1. Presence of other co morbid conditions that can contribute to gait dysfunction (orthopedic, rheumatologic, cardiac, other)
2. Presence of freezing of gait (FOG) ONLY in medications ON state
3. Presence of freezing of gait (FOG) ONLY in medications OFF state
4. Presence of significant cognitive dysfunction as determined by Montreal Cognitive Assessment (MoCA) <20
5. Presence of clinically significant depression as determined by geriatric depression scale (GDS)- 15>5
6. Presence of clinically significant hallucinations
7. Inability to sign informed consent
8. Participation in the physical therapy aimed at management of PD for the duration of the study (PT for orthopedic issues will be allowed)
9. Contraindications for use of Amantadine ( prior history of allergic reaction, history of known renal insufficiency with Cr > 2)
10. If female, be pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a total of 3 participants enrolled into the study. All 3 participants were randomized to receive either Amantadine or Placebo and crossed over after a washout period.
Groups:
- Amantadine, Then Placebo: Participants first received Amantadine 100 mg tablet orally once a day for one week, then two tablets orally twice a day for one week. After a washout period of 3 weeks, they then placebo tablet (matching Amantadine 100mg tablet) orally for 4 weeks.
- Placebo, Then Amantadine: Participants first received Placebo tablet (matching Amantadine 100 mg tablet) orally once a day for one week, then Amantadine placebo two tablets orally twice a day for one week. After a washout period of 4 weeks, then they received Amantadine 100mg tablet orally for 4 weeks.
Period: Overall Study
Arm/Group | Amantadine, Then Placebo | Placebo, Then Amantadine
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amantadine Crossover to Placebo: For first 4 weeks of study Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day
  Amantadine: Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day. Amantadine will then be administered orally twice daily in the morning with breakfast and at noon with lunch (AM and NN).
  Crossover to Placebo (sugar pill) at week 7
- Placebo Crossover to Amantadine: For first 4 weeks of study, Placebo (sugar pill)
  Crossover to Amantadine at week 7 Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day
  Amantadine: Amantadine 100mg daily, for a week, if it is tolerated Amantadine will increase to 1 tab twice a day. Amantadine will then be administered orally twice daily in the morning with breakfast and at noon with lunch (AM and NN).
- Total: Total of all reporting groups
Arm/Group | Amantadine Crossover to Placebo | Placebo Crossover to Amantadine | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Timed Up and Go (TUG) - ON Usual Medication
Description: This is a walking assessment. The subject will begin in the seated position, stand up, walk 7 meters, turn around, and sit back down. The entire process from leaving the chair to returning to the chair will be timed. Also, the Timed Up and Go (TUG) will be done both in the ON and OFF states.
Time Frame: Baseline, change at 4 weeks
Population: participants who could complete the task. Note: for the 2 participants who were tested while on placebo, one did not complete baseline, and one did not complete week 4, so a change could not be computed.
Measure: Median (Full Range); unit: seconds
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 3 | 1
seconds
  Baseline | 16.7 [15.86 to 18.16] | 17.4 [17.4 to 17.4]
  Change at 4 weeks: number analyzed (Participants) | 3 | 0
  Change at 4 weeks | 0.04 [-0.8 to 1.45] |

2. Primary Outcome: Timed Up and Go (TUG) - OFF Usual Medication
Description: as for outcome 1
Time Frame: Baseline, change at 4 weeks
Population: participants who could complete the task.
Measure: Median (Full Range); unit: seconds
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 2 | 2
seconds
  Baseline | 23 [20 to 24] | 19.5 [17 to 22]
  Change at 4 weeks | -3.5 [-4.3 to -2.7] | 8.6 [-0.2 to 17.5]

3. Secondary Outcome: Modified Timed Up and Go (mTUG)
Description: The subject sits in the chair approximately 3 1/2 meters away from doorway with the door closed. Subject then stands up and walks one meter to a 40cm X 40cm box taped on the floor. Within the box the patient turns clockwise (360 degrees), then turns counterclockwise (360 degrees). Walk to open the door and walk through the doorway, turn around and return to the chair. Modified Timed Up and Go (mTUG) completed in three components including walking the course without additional tasks, carrying a tray with a cup of water, and counting backwards from 100, in both ON and OFF state.
Time Frame: Baseline, change in 4 weeks
Population: participants who completed task
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 1 | 1
seconds
  Baseline - ON | 14 (0) | 16 (0)
  change in 4 weeks - ON | 1 (0) | -1 (0)
  Baseline - OFF | 16 (0) | 20 (0)
  change in 4 weeks - OFF | 2 (0) | 1 (0)

4. Secondary Outcome: Analysis of Motor Functioning Using the Parkinson's Home Diaries
Description: Subject will record motor activity as OFF, ON (mobility improved) or asleep on the diary every half hour for two days. Subjects further define ON time according to dyskinesia categories "none", "non-troublesome" or "troublesome." The home diaries are used as an evaluation measure of the intervention by assessing the change in off time and change in on time with troublesome dyskinesia. The difference in time experiencing dyskinesia while ON meds relative to the time OFF meds at baseline and at 4 weeks is compared.
Time Frame: Baseline, change in 4 weeks
Population: patients who report being ON and OFF medication and experience dyskinesia under either condition at baseline and after 4 weeks of either Amantadine or Placebo.
  NOTE: only one patient reported both dyskinesia at baseline and 4 weeks and only under the placebo condition. Others did not report any OFF time, so the difference could not be calculated.
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 1 | 1
minutes
  Baseline | 90 (0) | 150 (0)
  Change at 4 weeks: number analyzed (Participants) | 0 | 1
  Change at 4 weeks |  | 450 (0)

5. Secondary Outcome: Freezing of Gait Questionnaire
Description: A questionnaire that is used to assess the likelihood of the subject freezing in a number of different scenarios.
  0=No freezing of gait to 24=severe freezing of gait
Time Frame: Baseline, change in 4 weeks
Population: Participants who completed questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline | 10 [9 to 17] | 15 [13 to 17]
  Change at 4 weeks | -2 [-7 to 3] | 1 [-1 to 3]

6. Secondary Outcome: Clinical Global Impression (CGI)
Description: Global Improvement is the second scale in the clinical global impression (CGI). Total overall improvement is judged by whether or not, in the judgment of the assessor, the improvement is entirely due to the drug treatment. It is also a 1-7 point weighted scale, going from "very much improved" (1) to "very much worse" (7). A zero score is assigned if the score is not assessed.
Time Frame: 4 weeks
Population: number completing study up to assessment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 2 [2 to 6] | 4.5 [4 to 5]

7. Secondary Outcome: Parkinson's Disease Questionnaire-39 (PDQ-39)
Description: The Parkinson's Disease Questionnaire-39 (PDQ39) is a copyrighted instrument to assess symptoms of Parkinson's disease (PD) with 39 questions relating to mobility, activities of daily living, emotional well-being, social support, cognition, communication and bodily discomfort. The test asks subjects to rate each question regarding their Parkinson's disease symptoms over the past month. (range 0 to 100, lower scores reflect better quality of life)
Time Frame: Baseline, week 4
Population: Participants completing questionnaire
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 38 [32 to 43] |
  Week 4: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Gait Analysis Testing
Description: Use of an accelerometer such as Motorola Droid and wireless acceleration sensors to record gait parameters step time, walking speed, and cadence during the timed up and go (TUG) and modified timed up and go (mTUG) components. The sensors will be attached to the subject's legs and trunk using Velcro straps. The accelerometer will be held or clipped onto the subject in order to measure his or her acceleration. This is done within clinic and during the visit time.
Time Frame: Baseline, week 4, week 7, week 11
Population: No data was collected from the portable devices that were used.
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: A questionnaire used to discriminate between Parkinson Disease (PD) patients with fatigue and those without fatigue. Range 9 to 63, higher scores indicate greater fatigue severity.
Time Frame: Baseline, change in 4 weeks
Population: Participants who completed questionnaire
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline | 27 [13 to 32] | 26 [12 to 40]
  change in 4 weeks | 1.5 [0 to 3] | -5 [-10 to 0]

10. Secondary Outcome: Number Who Completed Medication as Randomized
Description: Tolerability analysis as determined by the number of subjects completing each arm of the study.
Time Frame: week 4
Population: participants who completed study to time of assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

11. Secondary Outcome: Number of Participants With Drug Safety Reports
Description: Analyzing the safety of the medication, Amantadine. Data regarding the medication will be collected from the patient on each visit including any adverse events since the last visit, frequency and severity of falls. This is done in order to determine the safety of Amantadine.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Amantadine: Participants during Amantadine 100 mg tablet orally once a day for one week, then two tablets orally twice a day for one week.
- Placebo: Participants during Placebo tablet (matching Amantadine 100 mg tablet)
Arm/Group | Amantadine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No